CLINICAL TRIAL: NCT00001638
Title: Cardiovascular Magnetic Resonance Imaging
Brief Title: Magnetic Resonance Imaging of the Blood Vessels of the Heart
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970204; 97-H-0204
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2009-08-04

CONDITIONS: Heart Disease
Keywords: Echocardiography; Heart; Gadolinium; Dobutamine; Toxicity; Adverse Events; Myocardial Infarction; Myocardial Viability; Myocardial Perfusion; Myocardial Function; Cardiovascular Disease
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction; Cardiovascular Diseases

SUMMARY:
This study is directed at evaluating patients with "myocardial ischemia" or poor blood supply to the heart muscle due to coronary artery disease. The major objective of this study is to determine the level of safety and effectiveness of magnetic resonance imaging at diagnosing coronary artery disease.

In addition, this study will allow researchers at the National Institutes of Health to see a broad spectrum of disease, preserve clinical skills, and stimulate future ideas for clinical research....

DETAILED DESCRIPTION:
This is a teaching protocol. It is in a format for training physicians in the laboratory in cardiovascular MRI techniques necessary for our research protocols. It helps provide experience necessary to develop and maintain our clinical expertise with cardiovascular MRI methods. It also provides physicians in the region access to this technology.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for All Arms of the Protocol

1. Known or suspected cardiovascular disease.
2. 18 years of age and older.
3. Able to provide informed consent.

Exclusion Criteria for All Arms of the Protocol:

Patients with a contraindication to MRI scanning will be excluded. These contraindications include patients with the following devices:

1. Central nervous system aneurysm clips
2. Implanted neural stimulator
3. Implanted cardiac pacemaker or defibrillator
4. Cochlear implant
5. Ocular foreign body (e.g. metal shavings)
6. Implanted insulin pump
7. Metal shrapnel or bullet.

In addition the following patient groups will be excluded:

1. Pregnant women (Patients who are uncertain as to whether they are pregnant will be required to have a screening urine or blood pregnancy test)
2. Patients with symptoms of myocardial ischemia occurring despite maximally tolerated doses of oral antianginal therapy and intravenous nitroglycerin

Furthermore, the following patient groups will be excluded from studies involving the administration of MRI contrast agents:

1. lactating women unless they are willing to discard breast milk for 24 hours
2. renal disease (estimated glomerular filtration rate [eGFR] less than 30 ml/min/1.73 m(2) body surface area)

The eGFR will be used to estimate renal function if reported by the laboratory. Otherwise, estimated glomerular filtration rate (eGFR) can be based on the Modification of Diet in Renal Disease (MDRD) study equation (see below) in subjects with stable renal function. This formula is not applicable to patients with acute renal insufficiency:

eGFR (ml/min/l.73 m(2))= 175 x (serum creatinine)-l.l54 x (age)-0.203 x 0.742 (if the subject is female) x 1.212 (if the subject is black)

Additional Exclusion Criteria for Dobutamine MRI

1. Myocardial infarction within 48 hours.
2. Uncontrolled heart failure
3. Severe hypertension (SBP greater than 200, DBP greater than 110)
4. Atrial fibrillation
5. Ventricular tachycardia
6. Frequent PVC's (more than 1 every 10 heart beats or nonsustained ventricular tachycardia (greater than 4)
7. Patients with narrow angle glaucoma or known or suspected severe bladder outlet obstruction due to prostatic hypertrophy will not receive atropine

Additional Exclusion Criteria for Vasodilator Stress MRI

1. Myocardial infarction within 48 hours.
2. Patients that are not considered medically stable by their physician (for example, severe heart failure that makes it difficult to breathe while lying flat or severe problems with heart rhythms).
3. Patients with 2nd or 3rd degree heart block are excluded from receiving the medicine adenosine (abnormalities that can be seen on your ECG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2916 (Actual)
Dates: Start 1997-09-29; Primary Completion 2009-08-03 (Actual); Study Completion 2009-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Frank JA, Mattay VS, Duyn J, Sobering G, Barrios FA, Zigun J, Sexton R, Kwok P, Woo J, Moonen C, et al. Measurement of relative cerebral blood volume changes with visual stimulation by 'double-dose' gadopentetate-dimeglumine-enhanced dynamic magnetic resonance imaging. Invest Radiol. 1994 Jun;29 Suppl 2:S157-60. doi: 10.1097/00004424-199406001-00052. No abstract available. PMID 7928216
- [Background] Mattay VS, Weinberger DR, Barrios FA, Sobering GS, Kotrla KJ, van Gelderen P, Duyn JH, Sexton RH, Moonen CT, Frank JA. Brain mapping with functional MR imaging: comparison of gradient-echo--based exogenous and endogenous contrast techniques. Radiology. 1995 Mar;194(3):687-91. doi: 10.1148/radiology.194.3.7862963.
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423